CLINICAL TRIAL: NCT07232927
Title: Evaluation of Hemostatic Agents in Partial Nephrectomy: A Prospective Randomized Trial
Brief Title: Evaluation of Hemostatic Agents in Partial Nephrectomy
Acronym: HEMOSTA-PN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Cagri Akpinar, assistant professor of urology, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: İ3-191-20
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Partial Nephrectomy; Hemostatic Agents; Localized Renal Cell Carcinoma
Keywords: Partial nephrectomy; Renal cell carcinoma; Hemostatic agents; FloSeal; Surgicel; Hemorrhage; Urinary leakage
MeSH Terms: conditions — Carcinoma, Renal Cell; Hemorrhage | interventions — Sutures; FloSeal Matrix; Surgicel

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, single-center, three-arm, parallel assignment clinical trial comparing standard parenchymal suturing (Group A), suturing with FloSeal® (Group B), and suturing with Surgicel® (Group C) during partial nephrectomy for localized renal tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - Suturing Only (Active Comparator): Standard parenchymal suturing technique without use of adjunctive hemostatic material.
  Interventions: Procedure: Standard Parenchymal Suturing
- Group B - Suturing + FloSeal® (Experimental): Parenchymal suturing performed with adjunctive application of gelatin-thrombin matrix (FloSeal®).
  Interventions: Procedure: Suturing with FloSeal®
- Group C - Suturing + Surgicel® (Experimental): Parenchymal suturing performed with adjunctive use of oxidized regenerated cellulose (Surgicel®).
  Interventions: Procedure: Suturing with Surgicel®

INTERVENTIONS:
Procedure: Standard Parenchymal Suturing — Standard parenchymal suturing technique performed during partial nephrectomy without the use of adjunctive hemostatic materials. Serves as the control arm in the study.
  Arms: Group A - Suturing Only
Procedure: Suturing with FloSeal® — Partial nephrectomy performed with parenchymal suturing combined with gelatin-thrombin matrix (FloSeal®) as an adjunctive hemostatic agent.
  Arms: Group B - Suturing + FloSeal®
Procedure: Suturing with Surgicel® — Partial nephrectomy performed with parenchymal suturing combined with oxidized regenerated cellulose (Surgicel®) as an adjunctive hemostatic agent.
  Arms: Group C - Suturing + Surgicel®

SUMMARY:
This prospective randomized study aims to evaluate the effect of adjunctive hemostatic agents (FloSeal® and Surgicel®) on perioperative outcomes in patients undergoing partial nephrectomy for localized renal tumors. A total of 150 patients were randomized into three groups: standard parenchymal suturing (Group A), suturing with FloSeal® (Group B), and suturing with Surgicel® (Group C). The study primarily investigates whether hemostatic agents reduce postoperative hemorrhage, urinary leakage, and positive surgical margin rates. Secondary outcomes include renal function change, operative and ischemia times, estimated blood loss, and hospital stay. All surgeries were performed by a single experienced surgeon at Ankara University Urology Department between January 2023 and December 2024.

DETAILED DESCRIPTION:
Partial nephrectomy (PN) is the standard surgical treatment for localized renal tumors, providing oncologic efficacy comparable to radical nephrectomy while preserving renal function. Despite technological advances, hemorrhage and urinary leakage remain major perioperative challenges. Various hemostatic agents have been introduced to improve intraoperative hemostasis and collecting system closure, including gelatin-thrombin matrices (FloSeal®) and oxidized regenerated cellulose (Surgicel®). However, the true clinical value of these agents remains controversial due to limited high-quality evidence.

This prospective, randomized, single-center trial was conducted at Ankara University Faculty of Medicine, Department of Urology. The study enrolled 150 patients with localized renal masses (clinical stage T1a-T1b) scheduled for partial nephrectomy between January 2023 and December 2024. Patients were randomized equally into three groups: Group A (suturing only), Group B (suturing with FloSeal®), and Group C (suturing with Surgicel®). All surgeries were performed by a single experienced urologic surgeon using open, laparoscopic, or robotic approaches according to tumor complexity and patient preference.

The primary endpoints were the incidence of clinically significant postoperative hemorrhage requiring transfusion, urinary leakage/fistula, and oncologic safety assessed by positive surgical margins. Secondary outcomes included operative and ischemia times, estimated blood loss, postoperative renal function, and length of hospital stay. Statistical analyses included ANOVA, chi-square, logistic regression, and ROC curve analyses to identify predictors of perioperative complications and surgical margin positivity.

This study provides prospective evidence that adjunctive hemostatic agents do not significantly reduce postoperative hemorrhage or urinary leakage rates and do not influence oncologic safety. Perioperative outcomes are mainly determined by tumor and surgical factors rather than the use of hemostatic materials.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Diagnosed with localized renal mass (clinical stage T1a-T1b) suitable for partial nephrectomy.
* Adequate preoperative renal function to undergo surgery.
* Signed informed consent obtained prior to study enrollment.
* Undergoing open, laparoscopic, or robotic partial nephrectomy performed by the same experienced surgeon.

Exclusion Criteria:

* Patients with solitary kidney or bilateral renal tumors.
* History of previous renal surgery on the same kidney.
* Evidence of metastatic disease or locally advanced (≥T2) renal tumors.
* Coagulopathy, bleeding disorders, or ongoing anticoagulant therapy that cannot be discontinued.
* Active urinary tract infection or systemic infection.
* Known allergy or hypersensitivity to gelatin or oxidized cellulose components.
* Patients who decline participation or withdraw consent.
* Incomplete perioperative data or loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically significant postoperative hemorrhage requiring blood transfusion | From postoperative Day 0 through postoperative Day 30
  Presence of postoperative bleeding requiring blood transfusion, radiologic, or surgical intervention, recorded according to standardized clinical criteria.
Incidence of postoperative urinary leakage or fistula | From postoperative Day 0 through postoperative Day 30
  Detection of urinary leakage based on drain creatinine measurement or radiologic evidence of fistula following partial nephrectomy.
Rate of positive surgical margins | At pathological assessment (Day of surgery)
  Pathologic assessment of surgical margins on resected tumor specimens to evaluate oncologic safety.

SECONDARY OUTCOMES:
Mean operative time and warm ischemia time | Intraoperative (Day of surgery)
  Duration of surgery (skin-to-skin time) and warm ischemia time measured intraoperatively in minutes.
Estimated blood loss during surgery | Intraoperative (Day of surgery)
  Total blood loss recorded by anesthesia team and surgical staff.
Change in postoperative renal function (serum creatinine and eGFR) | Preoperative (1 day before surgery) and postoperative Day 30
  Comparison of preoperative and postoperative serum creatinine and eGFR values to assess renal function preservation.
Postoperative hospital stay | From postoperative Day 0 until discharge, assessed for up to 30 days.
  Number of days from operation until hospital discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Medicine, Department of Urology, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Campbell SC, Novick AC, Belldegrun A, Blute ML, Chow GK, Derweesh IH, Faraday MM, Kaouk JH, Leveillee RJ, Matin SF, Russo P, Uzzo RG; Practice Guidelines Committee of the American Urological Association. Guideline for management of the clinical T1 renal mass. J Urol. 2009 Oct;182(4):1271-9. doi: 10.1016/j.juro.2009.07.004. Epub 2009 Aug 14. No abstract available. PMID 19683266
- [Result] Di Maida F, Campi R, Lane BR, De Cobelli O, Sanguedolce F, Hatzichristodoulou G, Antonelli A, Grosso AA, Noyes S, Rodriguez-Faba O, Keeley FX, Langenhuijsen J, Musi G, Klatte T, Roscigno M, Akdogan B, Furlan M, Simeone C, Karakoyunlu N, Marszalek M, Capitanio U, Volpe A, Brookman-May S, Gschwend JE, Smaldone MC, Uzzo RG, Kutikov A, Minervini A, Sib International Consortium. Predictors of Positive Surgical Margins after Robot-Assisted Partial Nephrectomy for Localized Renal Tumors: Insights from a Large Multicenter International Prospective Observational Project (The Surface-Intermediate-Base Margin Score Consortium). J Clin Med. 2022 Mar 23;11(7):1765. doi: 10.3390/jcm11071765. PMID 35407375
- [Result] Ljungberg B, Albiges L, Abu-Ghanem Y, Bedke J, Capitanio U, Dabestani S, Fernandez-Pello S, Giles RH, Hofmann F, Hora M, Klatte T, Kuusk T, Lam TB, Marconi L, Powles T, Tahbaz R, Volpe A, Bex A. European Association of Urology Guidelines on Renal Cell Carcinoma: The 2022 Update. Eur Urol. 2022 Oct;82(4):399-410. doi: 10.1016/j.eururo.2022.03.006. Epub 2022 Mar 26. PMID 35346519
- [Result] Zargar H, Khalifeh A, Autorino R, Akca O, Brandao LF, Laydner H, Krishnan J, Samarasekera D, Haber GP, Stein RJ, Kaouk JH. Urine leak in minimally invasive partial nephrectomy: analysis of risk factors and role of intraoperative ureteral catheterization. Int Braz J Urol. 2014 Nov-Dec;40(6):763-71. doi: 10.1590/S1677-5538.IBJU.2014.06.07. PMID 25615258
- [Result] Erlich T, Abu-Ghanem Y, Ramon J, Mor Y, Rosenzweig B, Dotan Z. Postoperative Urinary Leakage Following Partial Nephrectomy for Renal Mass: Risk Factors and a Proposed Algorithm for the Diagnosis and Management. Scand J Surg. 2017 Jun;106(2):139-144. doi: 10.1177/1457496916659225. Epub 2016 Jul 18. PMID 27431979
- [Result] Kola O, Smigelski M, Nagpal S, Gogaj R, Taneja SS, Wysock JS, Huang WC. Urine leak and vascular complications following robotic partial nephrectomy: a contemporary single-center experience. J Robot Surg. 2024 Oct 29;18(1):387. doi: 10.1007/s11701-024-02096-1. PMID 39470887
- [Result] Maurice MJ, Ramirez D, Kara O, Malkoc E, Nelson RJ, Caputo PA, Kaouk JH. Omission of Hemostatic Agents During Robotic Partial Nephrectomy Does Not Increase Postoperative Bleeding Risk. J Endourol. 2016 Aug;30(8):877-83. doi: 10.1089/end.2016.0192. PMID 27279548
- [Result] Basu S, Khan IA, Das RK, Dey RK, Khan D, Agarwal V. RENAL nephrometry score: Predicting perioperative outcomes following open partial nephrectomy. Urol Ann. 2019 Apr-Jun;11(2):187-192. doi: 10.4103/UA.UA_93_18. PMID 31040606
- [Result] Abu-Ghanem Y, Dotan Z, Kaver I, Zilberman DE, Ramon J. The use of Haemostatic Agents does not impact the rate of hemorrhagic complications in patients undergoing partial nephrectomy for renal masses. Sci Rep. 2016 Aug 30;6:32376. doi: 10.1038/srep32376. PMID 27572274
- [Result] Aykan S, Temiz MZ, Ulus I, Yilmaz M, Gonultas S, Suzan S, Semercioz A, Muslumanoglu AY. The Use of Three Different Hemostatic Agents during Laparoscopic Partial Nephrectomy: A Comparison of Surgical and Early Renal Functional Outcomes. Eurasian J Med. 2019 Jun;51(2):160-164. doi: 10.5152/eurasianjmed.2018.18293. PMID 31258357
- [Result] Veccia A, Autorino R. Is there a relation between preserved renal function and oncological outcomes in patients undergoing partial nephrectomy for renal cell carcinoma? Ann Transl Med. 2018 Nov;6(Suppl 1):S88. doi: 10.21037/atm.2018.11.01. No abstract available. PMID 30613663
- [Result] Tonyali S, Koni A, Yazici S, Bilen CY. The Safety and Efficacy of Adjuvant Hemostatic Agents During Laparoscopic Nephron-Sparing Surgery: Comparison of Tachosil and Floseal Versus No Hemostatic Agents. Urol J. 2017 Jan 23;15(1):21-25. doi: 10.22037/uj.v0i0.4090. PMID 29277887
- [Result] Richter F, Schnorr D, Deger S, Trk I, Roigas J, Wille A, Loening SA. Improvement of hemostasis in open and laparoscopically performed partial nephrectomy using a gelatin matrix-thrombin tissue sealant (FloSeal). Urology. 2003 Jan;61(1):73-7. doi: 10.1016/s0090-4295(02)02143-x. PMID 12559270
- [Result] Gill IS, Ramani AP, Spaliviero M, Xu M, Finelli A, Kaouk JH, Desai MM. Improved hemostasis during laparoscopic partial nephrectomy using gelatin matrix thrombin sealant. Urology. 2005 Mar;65(3):463-6. doi: 10.1016/j.urology.2004.10.030. PMID 15780356
- [Result] Carrion DM, Y Gregorio SA, Rivas JG, Bazan AA, Sebastian JD, Martinez-Pineiro L. The role of hemostatic agents in preventing complications in laparoscopic partial nephrectomy. Cent European J Urol. 2017;70(4):362-367. doi: 10.5173/ceju.2017.1432. Epub 2017 Oct 17. PMID 29410886
- [Result] Shao IH, Lee CL, Lin YH, Wang HS, Chen MC, Chang YH, Sheng TW, Huang LK, Kan HC, Liu CY, Lin PH, Yu KJ, Chuang CK, Pang ST, Wu CT. Predicting hemorrhagic complications in robotic-assisted partial nephrectomy for renal tumors: simplifying risk assessment with tumor diameter and depth. J Robot Surg. 2025 Jul 10;19(1):368. doi: 10.1007/s11701-025-02537-5. PMID 40637905
- [Result] Blachman-Braun R, Patel M, Loebach L, Millan B, Saini J, Gurram S, Linehan WM, Ball MW. Urinary leak after partial nephrectomy: Insights from a cohort with hereditary, multifocal, and reoperative cases. Urol Oncol. 2025 Aug;43(8):470.e11-470.e18. doi: 10.1016/j.urolonc.2025.03.013. Epub 2025 Apr 2. PMID 40180849
- [Result] Ryan J, MacCraith E, Davis NF, McLornan L. A systematic management algorithm for perioperative complications after robotic assisted partial nephrectomy. Can Urol Assoc J. 2019 Nov;13(11):E371-E376. doi: 10.5489/cuaj.5750. PMID 30817286
- [Result] Peyton CC, Hajiran A, Morgan K, Azizi M, Tang D, Chipollini J, Gilbert SM, Poch M, Sexton WJ, Spiess PE. Urinary leak following partial nephrectomy: a contemporary review of 975 cases. Can J Urol. 2020 Feb;27(1):10118-10124. PMID 32065869
- [Result] Li KP, Chen SY, Wang CY, Yang L. Comparison between minimally invasive partial nephrectomy and open partial nephrectomy for complex renal tumors: a systematic review and meta-analysis. Int J Surg. 2023 Jun 1;109(6):1769-1782. doi: 10.1097/JS9.0000000000000397. PMID 37094827
- [Result] Capitanio U, Terrone C, Antonelli A, Minervini A, Volpe A, Furlan M, Matloob R, Regis F, Fiori C, Porpiglia F, Di Trapani E, Zacchero M, Serni S, Salonia A, Carini M, Simeone C, Montorsi F, Bertini R. Nephron-sparing techniques independently decrease the risk of cardiovascular events relative to radical nephrectomy in patients with a T1a-T1b renal mass and normal preoperative renal function. Eur Urol. 2015 Apr;67(4):683-9. doi: 10.1016/j.eururo.2014.09.027. Epub 2014 Oct 3. PMID 25282367
- [Result] Cao Y, Cui Y, Li R, Tang X, Lin C, Yang X, Liu J, Zhao Q, Ma J, de Oliveira Paludo A, Schmeusser BN, Wang S, Du P. Comparing the long-term prognosis and renal function changes of partial nephrectomy (PN) and radical nephrectomy (RN) in T1 stage renal cell carcinoma patients. Transl Androl Urol. 2025 Mar 30;14(3):740-750. doi: 10.21037/tau-2025-136. Epub 2025 Mar 26. PMID 40226071